CLINICAL TRIAL: NCT00963118
Title: Bioactive Plant Foods: Effects on Functional Bioavailability and Genomic Stability
Acronym: Biogreen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: National Academy of Agricultural science, Korea (Unknown); Sungkyunkwan University (Other)
Responsible Party: Kyung-Jin Yeum, Tufts university
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: FRGN52
Record Dates: First submitted 2009-08-20; First posted 2009-08-21 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Metabolic Syndrome
Keywords: Angelica keiskei; Glycine max; metabolic syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- placebo (Placebo Comparator): Rice powder based nutrition bar
  Interventions: Dietary Supplement: plant based nutrition bar
- Angelica keiskei (Experimental): Angelica keiskei (green leafy vegetable) based nutrition bar
  Interventions: Dietary Supplement: plant based nutrition bar
- Glycine max (Experimental): Glycine max (black soybeans) based nutrition bar
  Interventions: Dietary Supplement: plant based nutrition bar
- Angelica keiskei + Glycine max (Experimental): Angelica keiskei (green leafy vegetable) and glycine max (black soybeans) based nutrition bar
  Interventions: Dietary Supplement: plant based nutrition bar

INTERVENTIONS:
Dietary Supplement: plant based nutrition bar — Nutrition bars made from Angelica keiskei (5g), glycine max (5g), Angelica keiskei (2.5g) + Glycine max (2.5g) or rice powder (12g) will be supplemented twice/day for 4 wks.

SUMMARY:
To achieve optimal health and to reduce the risk of age-related chronic diseases through an easily achievable dietary modification not achievable by the limited mixture of antioxidant supplements in older subjects, the investigators will focus their attention on the biological functions of bioactive plant food (Angelica keiskei and/or Glycine max) and its effect on genomic stability using noble assays.

The investigators propose to study the ability of bioactive plant-based food (Nutrition bar made from Angelica keiskei and/or Glycine max) to 1) exert biological functions: increase total antioxidant performance, decrease oxidative stress in vivo, and 2) affect genomic stability: decrease DNA damage and modify DNA methylation. The investigators hypothesize that bioactive plant food (green leafy vegetable power, and/or black bean power) will exert biological functions and affect genomic stability far more efficiently than the limited mixture of purified antioxidant supplements in the vulnerable population, older subjects (> 50 years, men and postmenopausal women) with and without metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria: healthy control group (n=20)

1. Age: over 50 years old
2. Female subjects must be post-menopausal
3. BMI: 18.5 - 30, waist/hip ratio < 0.9 for men, < 0.85 for women
4. TG<150 mg/dL (1.7 mmol/L) and no medication for TG
5. Total cholesterol < 200 mg /dL (5.18 mmol/L) and no medication for cholesterol
6. Blood pressure: SBP < 130 mmHg and DBP < 85 mmHg and no hypertensive medication
7. Plasma glucose: fasting blood glucose < 100 mg/dL (5.6 mmol/L) and no diabetes medication

Inclusion Criteria: Metabolic syndrome (n=40)

1. Age: over 50 years old
2. BMI: > 30 or waist/hip ratio > 0.9 for men, > 0.85 for women
3. Plus any two of the following four factors:

   * TG: 150-400 mg/dL (1.7 - 4.52 mmol/L) and/or medication for TG
   * HDL cholesterol: <40 mg /dL (1.03 mmol/L) for men, <50 mg/dL (1.29 mmol/L) for women and/or medication for cholesterol
   * Blood pressure: SBP, 130-160 mmHg and/or DBP 85-95 mmHg and/or antihypertensive medication
   * Plasma glucose: fasting blood glucose 100-125 mg/dL (5.55- 6.94 mmol/L) and no diabetes medication

Exclusion Criteria:

1. Study participants will be screened for normal hematologic parameters, normal serum albumin, normal liver function, normal kidney function, absence of fat malabsorption.
2. Subjects with a history of kidney stones, active small bowel disease or resection, atrophic gastritis, insulin-requiring diabetes, alcoholism, pancreatic disease, or bleeding disorders will be excluded from the study.
3. Exogenous hormone users will be excluded from the study.
4. Moreover, subjects will be non-smokers and will not have taken vitamin or carotenoid supplements for at least 6 weeks prior to the study and throughout the study for both healthy subjects and subjects with metabolic syndrome.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-06; Primary Completion 2010-07 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
plasma total antioxidant performance, DNA damage and DNA methylation | baseline, 2 & 4 wks after supplementation

SECONDARY OUTCOMES:
hydrophilic and lipophilic antioxidant nutrients (carotenoids, tocopherols, ascorbic acid and uric acid) | Baseline, 2 & 4 wks after supplementation

CONTACTS AND LOCATIONS:
Locations (1):
- Jean Mayer USDA-Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States